CLINICAL TRIAL: NCT04588389
Title: Comparison of Quadratus Lumborum Block With Medical Management for Pain Control After Lumbar Spine Fusion Surgery
Brief Title: Comparison of Quadratus Lumborum Block Types
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: PI left the institution. Decision made to close the study.
Sponsor: University of Massachusetts, Worcester (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: H00016236
Record Dates: First submitted 2020-09-30; First posted 2020-10-19 (Actual); Results first posted 2025-07-28 (Actual); Last update posted 2025-07-28 (Actual); Status verified 2025-07

CONDITIONS: Pain; Opioid Use; Lumbar Disc Herniation
Keywords: Lumbar Spine; Nerve Block; Opioid Use; Pain
MeSH Terms: conditions — Pain; Intervertebral Disc Displacement | interventions — Lidocaine; Standard of Care

STUDY DESIGN:
Intervention Model Description: We will randomize 10 patients into one of three groups for a total of 30 patients. Each patient will be longitudinally followed until discharge.
Who Masked: Participant, Outcomes Assessor
Masking Description: For the blinding purposes, the patients will be told that there are two possible sites at which they will receive the block. The sites will be either in the operating room before you wake up from anesthesia or in the post-anesthesia care unit (PACU). The patients on the medical management group will be told that they have received their block before recovering from anesthesia, the PACU nurse will be told the same as well to make him or her blinded as a pain assessor.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (3):
- Group 1 Standard of Care (Active Comparator): Group I will receive the standard of care multimodal pharmacological management.
  Interventions: Drug: Multimodal Pharmacological Management
- Group 2 Standard of Care + Quadratus Lumborum Block II (Experimental): Group II will receive standard of care multimodal pharmacological management plus the Quadratus Lumborum II local anesthetic block.
  Interventions: Drug: Ropivacaine injection Location 1; Drug: Multimodal Pharmacological Management
- Group 3 Standard of Care + Quadratus Lumborum Block III (Experimental): Group III will receive standard of care multimodal pharmacological management plus the Quadratus Lumborum III local anesthetic block. We will measure opioid use, pain, and side effects in each patient.
  Interventions: Drug: Ropivacaine injection Location 2; Drug: Multimodal Pharmacological Management

INTERVENTIONS:
Drug: Ropivacaine injection Location 1 — Ropivacaine .5% and lidocaine 1% to the area behind the muscle Quadratus Lumborum location 1
  Other Names: Lidocaine
  Arms: Group 2 Standard of Care + Quadratus Lumborum Block II
Drug: Ropivacaine injection Location 2 — Ropivacaine .5% and lidocaine 1% to the area behind the muscle Quadratus Lumborum location 2
  Other Names: Lidocaine
  Arms: Group 3 Standard of Care + Quadratus Lumborum Block III
Drug: Multimodal Pharmacological Management — standard of care multimodal pharmacological management
  Other Names: Standard of Care

SUMMARY:
This study will compare the quality of analgesia and reduction of opioid use, between standard of care and two groups of local anesthetic blocks in different location in the quadratus lumborum plane, for postoperative pain control after lumbar spinal fusion and if it reduces opioid consumption.

DETAILED DESCRIPTION:
This study is a pilot study as part of planning for a larger randomized controlled trial. The study plans to enroll a total of 30 patients, with 10 patients randomly assigned in each group of the study. Group I will receive the standard of care multimodal pharmacological management. Group II will receive standard of care multimodal pharmacological management plus the Quadratus Lumborum II local anesthetic block. Group III will receive standard of care multimodal pharmacological management plus the Quadratus Lumborum III local anesthetic block. Measurements of opioid use, pain, and side effects will be recorded for each patient.

ELIGIBILITY:
Inclusion Criteria:

* Adult Patients undergoing lumbar spinal fusion surgery.
* Patients from 40-80 years.

Exclusion Criteria:

* Recent drug abuse
* History of illicit drug use
* Chronic pain patients not related to the back lesions.
* Opioid tolerant patients.
* Patients with any lower extremity weaknesses or deficits.
* Patients with American Society of Anesthesiologists (ASA) classification more than 3.
* Coagulopathy.
* Infection near or in the area of the block.
* Pregnant patients.
* Uncooperative patients who refuse care which directly effects research participation or clinical care.
* If the surgeon reports performing non-typical fusion.
* The presence of intraoperative complications like nerve injury or abnormal results of neuromonitoring and extensive dissection.
* Vulnerable populations (prisoner, mental impairment / dementia, pregnant, etc.)
* Subjects on chronic buprenorphine therapy (either for opioid replacement or pain control)

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2020-12-01 (Actual); Primary Completion 2021-05-14 (Actual); Study Completion 2021-05-14 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Eman Nada, MD, Principal Investigator — University of Massachusetts, Worcester; Alexander Chan, MD, Principal Investigator — University of Massachusetts, Worcester
Locations (1):
- UMASS Memorial Medical Center, Worcester, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No
There is no plan to share individual participant data with other researchers. However, results of the study will be shared through publication.

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Group 1 Standard of Care | Group 2 Standard of Care + Quadratus Lumborum Block II | Group 3 Standard of Care + Quadratus Lumborum Block III
Started | 2 | 4 | 3
Completed | 0 | 4 | 3
Not Completed | 2 | 0 | 0
Not completed — Issues with anesthesia during surgery | 2 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Per participant flow, 0 Group 1 participants are included in analysis population. The data from two patients in Group I was NOT collected because there was a protocol violation; one patient received Ketamine intraoperatively and the other patient received large amounts of local anesthetics in the wound.
Groups:
- Total: Total of all reporting groups
Arm/Group | Group 1 Standard of Care | Group 2 Standard of Care + Quadratus Lumborum Block II | Group 3 Standard of Care + Quadratus Lumborum Block III | Total
Number analyzed (Participants) | 0 | 4 | 3 | 7
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 0 | 2 | 0 | 2
  >=65 years | 0 | 2 | 3 | 5
Age, Continuous [Mean (Full Range); unit: years] |  | 63.75 [51 to 74] | 73 [69 to 76] | 67.71 [51 to 76]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female |  | 3 | 3 | 6
  Male |  | 1 | 0 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native |  | 0 | 0 | 0
  Asian |  | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander |  | 0 | 0 | 0
  Black or African American |  | 0 | 0 | 0
  White |  | 0 | 0 | 0
  More than one race |  | 0 | 0 | 0
  Unknown or Not Reported |  | 4 | 3 | 7
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 0 | 4 | 3 | 7

OUTCOME MEASURES:

1. Primary Outcome: Opioid Consumption
Description: Dose of the opioids consumed
Time Frame: 12 hours
Population: No data was collected on Participants in Group 1 and were excluded from analysis population as there were issues with anesthesia. One participant received a large amount of local anesthetics by surgeon and the other received ketamine in anesthesia.
Measure: Mean (Full Range); unit: morphine milligram equivalents
Arm/Group | Group 1 Standard of Care | Group 2 Standard of Care + Quadratus Lumborum Block II | Group 3 Standard of Care + Quadratus Lumborum Block III
Number analyzed (Participants) | 0 | 4 | 3
morphine milligram equivalents |  | 30 [7.5 to 37.5] | 17.5 [7.5 to 22.5]

2. Primary Outcome: Opioid Consumption
Description: Dose of the opioids consumed
Time Frame: 24 hours
Population: as for outcome 1
Measure: Mean (Full Range); unit: Morphine milligram equivalents
Arm/Group | Group 1 Standard of Care | Group 2 Standard of Care + Quadratus Lumborum Block II | Group 3 Standard of Care + Quadratus Lumborum Block III
Number analyzed (Participants) | 0 | 4 | 3
Morphine milligram equivalents |  | 31 [7.5 to 56.25] | 20 [15 to 37.5]

3. Primary Outcome: Opioid Consumption
Description: Dose of the opioids consumed
Time Frame: 36 hours
Population: as for outcome 1
Measure: Mean (Full Range); unit: Morphine milligram equivalents
Arm/Group | Group 1 Standard of Care | Group 2 Standard of Care + Quadratus Lumborum Block II | Group 3 Standard of Care + Quadratus Lumborum Block III
Number analyzed (Participants) | 0 | 4 | 3
Morphine milligram equivalents |  | 35.625 [15 to 52.5] | 20 [7.5 to 30]

4. Primary Outcome: Opioid Consumption
Description: Dose of the opioids consumed
Time Frame: 48 hours
Population: as for outcome 1
Measure: Mean (Full Range); unit: Morphine milligram equivalents
Arm/Group | Group 1 Standard of Care | Group 2 Standard of Care + Quadratus Lumborum Block II | Group 3 Standard of Care + Quadratus Lumborum Block III
Number analyzed (Participants) | 0 | 4 | 3
Morphine milligram equivalents |  | 31.875 [15 to 45] | 25 [15 to 30]

5. Secondary Outcome: Pain Scale
Description: Numerical Pain Scale Rating, likert scale of 0-10 with a 0 indicating absence of pain and 10 indicating worst pain imaginable.
Time Frame: 0 Hours
Population: as for outcome 1
Measure: Mean (Full Range); unit: score on a scale
Arm/Group | Group 1 Standard of Care | Group 2 Standard of Care + Quadratus Lumborum Block II | Group 3 Standard of Care + Quadratus Lumborum Block III
Number analyzed (Participants) | 0 | 4 | 3
score on a scale |  | 8 [5 to 10] | 3.67 [0 to 7]

6. Secondary Outcome: Pain Scale
Description: Numerical Pain Scale Rating of 0-10 with a 0 indicating absence of pain and 10 indicating worst pain imaginable.
Time Frame: 1 Hour
Population: as for outcome 1
Measure: Mean (Full Range); unit: score on a scale
Arm/Group | Group 1 Standard of Care | Group 2 Standard of Care + Quadratus Lumborum Block II | Group 3 Standard of Care + Quadratus Lumborum Block III
Number analyzed (Participants) | 0 | 4 | 3
score on a scale |  | 4.75 [3 to 8] | 2 [0 to 4]

7. Secondary Outcome: Pain Scale
Description: as for outcome 5
Time Frame: 6 Hours
Population: as for outcome 1
Measure: Mean (Full Range); unit: score on a scale
Arm/Group | Group 1 Standard of Care | Group 2 Standard of Care + Quadratus Lumborum Block II | Group 3 Standard of Care + Quadratus Lumborum Block III
Number analyzed (Participants) | 0 | 4 | 3
score on a scale |  | 5.25 [3 to 8] | 2.33 [0 to 4]

8. Secondary Outcome: Pain Scale
Description: as for outcome 5
Time Frame: 12 Hours
Population: as for outcome 1
Measure: Mean (Full Range); unit: score on a scale
Arm/Group | Group 1 Standard of Care | Group 2 Standard of Care + Quadratus Lumborum Block II | Group 3 Standard of Care + Quadratus Lumborum Block III
Number analyzed (Participants) | 0 | 4 | 3
score on a scale |  | 5.25 [4 to 8] | 5.33 [4 to 8]

9. Secondary Outcome: Pain Scale
Description: as for outcome 5
Time Frame: 18 Hours
Population: as for outcome 1
Measure: Mean (Full Range); unit: score on a scale
Arm/Group | Group 1 Standard of Care | Group 2 Standard of Care + Quadratus Lumborum Block II | Group 3 Standard of Care + Quadratus Lumborum Block III
Number analyzed (Participants) | 0 | 4 | 3
score on a scale |  | 6 [4 to 9] | 5.33 [3 to 8]

10. Secondary Outcome: Pain Scale
Description: as for outcome 5
Time Frame: 24 Hours
Population: as for outcome 1
Measure: Mean (Full Range); unit: score on a scale
Arm/Group | Group 1 Standard of Care | Group 2 Standard of Care + Quadratus Lumborum Block II | Group 3 Standard of Care + Quadratus Lumborum Block III
Number analyzed (Participants) | 0 | 4 | 3
score on a scale |  | 5.75 [4 to 7] | 4.67 [3 to 6]

11. Secondary Outcome: Pain Scale
Description: as for outcome 5
Time Frame: 30 Hours
Population: as for outcome 1
Measure: Mean (Full Range); unit: score on a scale
Arm/Group | Group 1 Standard of Care | Group 2 Standard of Care + Quadratus Lumborum Block II | Group 3 Standard of Care + Quadratus Lumborum Block III
Number analyzed (Participants) | 0 | 4 | 3
score on a scale |  | 4.75 [0 to 8] | 2.3 [0 to 5]

12. Secondary Outcome: Pain Scale
Description: as for outcome 5
Time Frame: 36 Hours
Population: as for outcome 1
Measure: Mean (Full Range); unit: score on a scale
Arm/Group | Group 1 Standard of Care | Group 2 Standard of Care + Quadratus Lumborum Block II | Group 3 Standard of Care + Quadratus Lumborum Block III
Number analyzed (Participants) | 0 | 4 | 3
score on a scale |  | 6.25 [4 to 9] | 6.33 [4 to 10]

13. Secondary Outcome: Pain Scale
Description: as for outcome 5
Time Frame: 42 Hours
Population: as for outcome 1
Measure: Mean (Full Range); unit: score on a scale
Arm/Group | Group 1 Standard of Care | Group 2 Standard of Care + Quadratus Lumborum Block II | Group 3 Standard of Care + Quadratus Lumborum Block III
Number analyzed (Participants) | 0 | 4 | 3
score on a scale |  | 5.25 [4 to 7] | 2 [0 to 6]

14. Secondary Outcome: Pain Scale
Description: as for outcome 5
Time Frame: 48 hours
Population: No data was collected on Participants in Group 1 and were excluded from analysis population as there were issues with anesthesia. One participant received a large amount of local anesthetics by surgeon and the other received ketamine in anesthesia.
  Not able to collect data on a Group 2 participant due to timing and discharge.
Measure: Mean (Full Range); unit: score on a scale
Arm/Group | Group 1 Standard of Care | Group 2 Standard of Care + Quadratus Lumborum Block II | Group 3 Standard of Care + Quadratus Lumborum Block III
Number analyzed (Participants) | 0 | 3 | 3
score on a scale |  | 6 [4 to 8] | 3.667 [3 to 4]

15. Secondary Outcome: Discharge Opioid Use
Description: The amount of left-over opioid pills at 2 weeks in the follow up visit.
Time Frame: 2 weeks
Population: as for outcome 1
Arm/Group | Group 1 Standard of Care | Group 2 Standard of Care + Quadratus Lumborum Block II | Group 3 Standard of Care + Quadratus Lumborum Block III
Number analyzed (Participants) | 0 | 0 | 0

16. Secondary Outcome: Number of Participants Experiencing Side Effects
Description: Number of Participants who experienced side effects.
Time Frame: Up to 1 week
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | Group 1 Standard of Care | Group 2 Standard of Care + Quadratus Lumborum Block II | Group 3 Standard of Care + Quadratus Lumborum Block III
Number analyzed (Participants) | 0 | 4 | 3
participants |  | 4 | 3

ADVERSE EVENTS:
Time Frame: 4 months, 14 days. This is equal to the specified time the study was conducted.
Arm/Group | Group 1 Standard of Care | Group 2 Standard of Care + Quadratus Lumborum Block II | Group 3 Standard of Care + Quadratus Lumborum Block III
All-Cause Mortality (participants affected / at risk) | 0/2 | 0/4 | 0/3
Serious Adverse Events (participants affected / at risk) | 0/2 | 0/4 | 0/3
Other Adverse Events (participants affected / at risk) | 0/2 | 0/4 | 0/3

LIMITATIONS AND CAVEATS:
Research project closed early due to departure of originating PI and despite departmental efforts, a new PI was not available to take over study. Study encountered coordination issues relative to Arm 1.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2018-09-17): https://cdn.clinicaltrials.gov/large-docs/89/NCT04588389/Prot_SAP_000.pdf
  • Informed Consent Form (2021-04-20): https://cdn.clinicaltrials.gov/large-docs/89/NCT04588389/ICF_002.pdf